CLINICAL TRIAL: NCT04477265
Title: Efficacy of of Pelvic Floor Muscle Training( PFMT ) With Surface Electromyographic Biofeedback and Medication in Women With Overactive Bladder
Brief Title: Efficacy of Biofeedback PFMT and Medication in Women With Overactive Bladder
Acronym: PFMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 105019 - F
Record Dates: First submitted 2020-06-15; First posted 2020-07-20 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2020-05

CONDITIONS: Overactive Bladder
Keywords: Overactive; drug only; exercise only; combination of drug and exercise
MeSH Terms: conditions — Urinary Bladder, Overactive; Motor Activity | interventions — Solifenacin Succinate

STUDY DESIGN:
Intervention Model Description: A total of 210 women with overactive bladder will be recruited and randomized to 3 arms: drug only, exercise only and combination arm.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- combination of drug and exercise (Experimental): Participant will be prescribed with oral medication in combination with biofeedback-assisted pelvic floor muscle training (PFMT) during the first month, participant will continue to have biofeedback assisted PFMT for another 2 months
  Interventions: Drug: Solifenacin Succinate 5mg/tab daily; Behavioral: biofeedback-assisted pelvic floor muscle training
- drug only (Active Comparator): Participant will be prescribed with oral medication for 3 months
  Interventions: Drug: Solifenacin Succinate 5mg/tab daily
- exercise only (Active Comparator): Participant will be doing biofeedback-assisted pelvic floor muscle training for 3 months
  Interventions: Behavioral: biofeedback-assisted pelvic floor muscle training

INTERVENTIONS:
Drug: Solifenacin Succinate 5mg/tab daily — participants will be taking oral medication for 3 months
  Other Names: Vesicare 5mg/tab daily
  Arms: combination of drug and exercise; drug only
Behavioral: biofeedback-assisted pelvic floor muscle training — participants will be doing biofeedback-assisted pelvic floor muscle training for 3 months
  Arms: combination of drug and exercise; exercise only

SUMMARY:
Medical treatment for overactive bladder is acceptable widely. However, the effect of drug treatment is different due to compliance and side effect of the drug. Biofeedback-assisted pelvic floor muscle training (PFMT) is the first line recommendation for overactive bladder. The slow effect of biofeedback-assisted pelvic floor muscle training leads to low motivation for continuous treatment and results in compliance difference. This slow effect also changes the degree of improvement in the treatment of overactive bladder. This study is designed to evaluate the efficacy of combination therapy for treatment of female overactive bladder.

DETAILED DESCRIPTION:
Participant will be prescribed with oral medication in combination with biofeedback-assisted pelvic floor muscle training (PFMT) for the first month. Participant will continue to have biofeedback assisted PFMT for another two months without oral medication. The investigators expected that combination therapy will improve the compliance and severity of symptoms in women with overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

1. overactivity bladder for more than 3 months
2. more then 20 year old,less then 85 year old and acceptable to receive vaginal examination
3. need to match schedule with the investigator's clinic for 5 times,followed by individual therapy, each takes about 30 to 60 minutes, a total of 12 weeks of pelvic floor muscle exercises

Exclusion Criteria:

1. Suffering from systemic neuromuscular diseases, such as stroke, spinal cord injury, peripheral neuropathy, etc.
2. Glaucoma
3. Kidney disease
4. Liver disease
5. Patients with cardiac rhythm devices.
6. Insufficient cognitive function, unable to cooperate with pelvic floor muscle exercises.
7. Women during pregnancy.
8. Maternity within six weeks after delivery

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
3-Day Voiding Diary | Baseline through study completion, an average of 12 weeks.
  to record urinary output, fluid consumed, and urinary leakage (if applicable) for 3 complete 24-hour periods (they do not have to be consecutive days).
Symptom Distress scale(SDS) | through study completion, an average of 12 weeks.
  the degree of discomfort from the specific symptoms being experienced, as perceived by the participants, consists of 23 items.The scale scored between 1 (best) and 5 (worst) .
change of electromyographic activity | through study completion, an average of 12 weeks.
  Electromyographic activity of the pelvic floor muscles (PFMs) and the synergistic abdominal muscles (SAMs) during each session of PFMT(µV)
King's Health Questionnaire (KHQ) | through study completion, an average of 12 weeks.
  KHQ has 3 parts consisting of 21 items. Part 1 contains general health perception and incontinence impact (one item each). Part 2 contains role limitations, physical limitations, social limitations (two items each), personal relationships, emotions (three items each) and sleep/energy (two items), severity measures (four items).Part 3 is considered as a single item and contains ten responses in relation to frequency, nocturia, urgency,urge, stress, intercourse incontinence, nocturnal enuresis,infections, pain, and difficulty in voiding. The 4 subscales scored between 1 (best) and 4 (worst) in part 1 and 2. The Symptom Severity scale is scored from 0 (best) to 3 (worst) in part 3 .
A five-item Self-Assessment of Treatment (SAT) | through study completion, an average of 12 weeks.
  to assess improvement and satisfaction with treatment, consists of 1 item. The scale scored between 1 (worst) and 5 (best ) .
A five-item Self-Assessment of Self-efficacy | through study completion, an average of 12 weeks.
  to assess motivation with PFMT, consists of 14 items.The scale scored between 1 (worst) and 6(best) .

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Yih Wu, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan